CLINICAL TRIAL: NCT04268680
Title: Perioperative Case Series: Qualitative Evaluation of Gait Cycle and Ground in Knee
Brief Title: Perioperative Case Series: Qualitative Evaluation of Gait Cycle and Ground in Knee Arthroplasty Patients
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: OpenGO
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-02

CONDITIONS: Gait, Unsteady
Keywords: gait cycle; knee arthroplasty; wearable insole
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gait analysis is a quick and powerful tool with a wide range of clinical applications in various fields. However, due to the expensive and highly specialized equipment required, gait studies are mostly limited to academic research centers and small sample sizes and no large-scale, randomized controlled trials have been performed. Several authors have proposed inexpensive accelerometer-based systems to remedy this situation. Through mathematic transformation they adequately measure step time and length. With these systems however only temporal spatial gait parameters can be recorded; kinetic gait parameters, such as ground reaction force, cannot be measured. As these kinetic parameters are important for clinical studies, especially in fracture and rehabilitation research different methods are needed. Its availability is mainly limited to research centers, conventional gait analysis is further hindered by its stationarity and that it only allows momentary views of the patient's gait in a confined research environment. Even smaller, wearable systems have to be attached to an external apparatus, or are limited by their battery capacity, data storage and other device specific factors. Furthermore, the use of these systems is at an early clinical stage and their full potential not yet developed. As most disease processes are continuous, tools with long-term, continuous measuring capabilities are needed. For this reason a new pressure-measuring insole with built in battery and data storage was developed in cooperation with the AO Foundation(AO Foundation, Davos, Switzerland). The system offers complete independence from any external measures for up to 4 weeks and monitors a patient step during this time.

The purpose of this pilot study is to investigate which how TKA arthroplasty may impact gait during early and medium term rehabilitation phase. This will be done through the use of the OpenGo Sensor Insole (Moticon GmbH).

DETAILED DESCRIPTION:
Advanced degenerative arthropathies of the knee ultimately manifest as pain and a loss of function leading to impaired gait and activity. Total knee arthroplasty (TKA) is a procedure that aim to eliminate pain, restore the function of the joint and ultimately improve the ability of the patient to move and live an active life. TotalKneeArthroplasty has a history of success, but as the orthopedic and healthcare sectors evolve, a greater level of scrutiny and expectation for success will be applied to surgeons and device makers alike. In response to these elevated levels of scrutiny and expectation more advanced methods will likely be required to better capture and understand how a TotalKneeArthroplasty impacts patient function both on an individual, patient by patient, basis as well as on device design and surgical technique basis.

The present study is aimed at performing a preliminary evaluation to provide:

More advanced insight into a patient's functional recovery and rehabilitation with the potential for phisician's to intervene earlier and with greater specificity to any challenges encountered by the patient Objective evidence of the quality and value of the intervention on an individualized basis. Study objectives Any change in gait as a result of arthroplasty and dynamics of gait recovery during acute recovery and rehabilitation timeframe. Outcome measures will be gait cycle and ground: foot interaction dynamics which will be observed longitudinally and compared to the healthy contralateral limb (ground: foot interaction dynamics) as well literature data (gait cycle).

Primary objective:Evaluation of gait cycle and ground in primary TotalKneeArthroplasty patients compared to the healthy contralateral limb.

Secondary objectives:Easy of use. Qualitative user (Phisician and patient) feedback on experience using and wearing the insoles Study design:This is, single arm, prospective, single center, pilot study to measure the pre-operative and post-operative gait and ground: foot interaction dynamics of 6 subjects who are undergoing TotalKneeArthroplasty .

Data that will be collected at baseline (pre-op) besides the standard clinical data (VisualAnalogueScale, KneeSocietyScore SatisfactionForm-12, Knee Injury and Osteoarthritis Outcome Score(KOOS)) include: gait and ground: foot interaction dynamics during a prescribed in clinic activity as well as during activities of daily living.

Data that will be collected about the clinical follow-up include: gait and ground: foot interaction dynamics during a prescribed in clinic activity as well as during activities of daily living; user feedback regarding their experience using and wearing the insoles.

Total study duration for study participants will be 6 months with follow-up visits planned at: daily until discharge, 1 week, 2 weeks, 3 weeks, 3 months and 6 months. Full enrollement is estimated to require 1 months, therefore the total study duration is expected to be 7 months.

Subjects will be included in 1 Italian site. Data and user feedback will be analyzed continuously as they become available throughout the study period.

Patients selection:Once a subject has completed the informed consent procedure and signed the Informed Consent Form, the PI or delegated study research staff can complete the screening process with the subject. All potential subjects who undergo the screening process will be documented on a Screening and Enrollment Log, on which reasons for exclusion from or denial to participate should be noted.

ELIGIBILITY:
Inclusion Criteria:

* primary TKA
* 45-75 years of age (included)
* skeletally mature
* willing and able to participate in required pre-op and follow-up visits at the investigational site and to complete study procedures and questionnaires
* consented to participating in the study by signing the IRB/EC approved informed consent form
* BMI <32

Exclusion Criteria:

* symptomatic/debilitating co-commitant arthropathy of non-operative joints (e.g. a TKA patient cannot have advanced arthritis of the contralateral knee or ipsilateral hip/ankle) that would impede or otherwise confuse the peri-operative measurement of gait.
* Significant comorbidities that would impede the patients ability to participate in standard recovery and rehabilitation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by degenerative gonarthrosis who need a TKA in one of the two Knees
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Perioperative Case Series: clinical evaluation of gait cycle and ground in Knee arthroplasty patients | baseline to 3 month
  Evaluation of gait cycle and ground in primary TKA patients compared to the healthy contralateral limb.

SECONDARY OUTCOMES:
Perioperative Case Series: qualitative evaluation of gait cycle and ground in Knee arthroplasty patients | baseline to 3 month
  Easy of use. Qualitative user (HCP and patient) feedback on experience using and wearing the insoles

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ulivi, Dr, Principal Investigator — IRCCS Istituto Ortopedico GaleazziMilano
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy